CLINICAL TRIAL: NCT00534183
Title: Metabolic Profile and Anthropometric Changes in Schizophrenia
Acronym: MetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Psychiatry, Ranchi, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CIPMETS001
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Metabolic Syndrome; Diabetes; Obesity
Keywords: Metabolic syndrome; Obesity; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Obesity | interventions — Olanzapine; Risperidone; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Olanzapine
  Interventions: Drug: Olanzapine
- 2 (Active Comparator): Risperidone
  Interventions: Drug: Risperidone
- 3 (Active Comparator): haloperidol
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Olanzapine — Olanzapine in dose range of 10-20mg
  Arms: 1
Drug: Risperidone — Risperidone 1-6mg
  Arms: 2
Drug: Haloperidol — Haloperidol 10-20mg
  Arms: 3

SUMMARY:
"No clinical differences will be found between the three antipsychotics under study - olanzapine, risperidone and haloperidol - on the patients' metabolic profile and weight. "

DETAILED DESCRIPTION:
we aimed to study the effects of antipsychotics, olanzapine, risperidone and haloperidol on development of metabolic syndrome in a drug naïve population suffering from first episode schizophrenia and compared it with a matched healthy control group. We also aimed to examine the prevalence of metabolic syndrome as defined by the two most widely accepted definitions, the ATP IIIA and the IDF.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years
* Diagnosis of schizophrenia
* Drug naive on admission

Exclusion Criteria:

* Other psychiatric co-morbidity
* History of severe physical illness
* Alcohol and substance abuse or dependence
* History of pre-existing diabetes or hypertension
* Family history of hypertension or diabetes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2006 (Actual)
Dates: Start 2006-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Study of metabolic profile | 6 weeks

SECONDARY OUTCOMES:
Study of obesity and diabetes | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sahoo Saddichha, DPM, Principal Investigator — Central Institute of Psychiatry
Locations (1):
- Central Institute of Psychiatry, Ranchi, India

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149
- [Derived] Saddichha S, Manjunatha N, Ameen S, Akhtar S. Effect of olanzapine, risperidone, and haloperidol treatment on weight and body mass index in first-episode schizophrenia patients in India: a randomized, double-blind, controlled, prospective study. J Clin Psychiatry. 2007 Nov;68(11):1793-8. doi: 10.4088/jcp.v68n1120. PMID 18052574